CLINICAL TRIAL: NCT03324100
Title: Crosstalk of Nasal Epithelium and Mucus in the Immune Response to Allergic Rhinitis: an Integrative Omics Approach to Measure Abundance Changes in Protein and RNA Expression
Brief Title: Integrative Omics Approach to Allergic Rhinitis
Acronym: IntegOmics
Status: Active, not recruiting | Type: Observational
Sponsor: Medical University of Graz (Other)
Collaborators: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Sponsor
Other Study IDs: IntegrativeOmics
Record Dates: First submitted 2017-10-20; First posted 2017-10-27 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Allergic Rhinitis Patients
- Healthy Controls

SUMMARY:
Nasal mucus and nasal epithelium are the first defense barriers against allergens. Various proteins are found in nasal mucus that play a role in allergic rhinitis and reflect immune response to allergen exposure. The difference in the proteomic profile of allergic rhinitis patients and healthy controls can give insight about how the response works and which proteins could lead to either enhanced immune reaction or to defense response like augmentation of epithelial integrity. It is also known that the airway epithelium plays a crucial role in the regulation of airway immune responses and inflammation. Gene expression profiling is widely used to analyses complex disease. For the airway epithelium gene expression profile in diseased and healthy state as well as in baseline and provoked state can clarify the mechanism of defense reactions and the course of inflammatory processes. Nasal mucus proteins as consequence of different gene expression can be seen as part of the end products of this complex mechanisms and interactions between allergens and the epithelium.

Nasal mucus proteins have different origins and production sites and gene expression does not necessarily result in functional metabolites. The aim of this proposed project is to try and analyze in a holistic proteomic approach the response to allergen on a genetic/genomic level from the nasal epithelium to protein/proteomic level in nasal mucus. This analysis gives us insight of how the different gene expression profiles result in a protein expression and further clarifies which proteins are directly originate from the epithelium and which are result of plasma exudation or underlie different regulatory processes.

From allergic rhinitis patients and healthy controls nasal mucus, nasal mucosa, and serum will be obtained. Nasal mucus will be collected with a special suction device equipped with a mucus trap from the middle meatus under endoscopic control without touching the mucosa. Nasal mucosa will be obtained through nasal brushes under local anesthesia and put into primary culture. Serum prepared from blood samples. Patients with grass or tree pollen allergy will be included and allergic state will be determined by skin prick tests and RAST (Radio-Allergo-Sorbent-test). The aimed for sample size will be 15 patients per group. Samples will be obtained in and out of pollen season. Allergic patients will fill out a symptom score and samples will be taken when symptoms are strong (in pollen season) and disappeared (out of pollen season). For healthy controls the time point of sample taking will be correlated to the allergic rhinitis patients to have a similar pollen exposure. Nasal mucus will be sent for Liquid Chromatography Tandem mass spectrometry for proteomic analysis and from nasal epithelial cells RNA will be isolated and send for Microarray analysis. By an integrative omics approach gene and protein expression will be correlated and cross talk between nasal mucus and epithelium will be analysed. The identification of key genes or gene clusters leads to further identification of key proteins or protein groups as biomarkers that could serve for novel therapeutic or diagnostic strategies in allergic rhinitis. The integrative omic approach downsizes the potential candidates since the focus lies on epithelial gene expression and their protein products and excludes proteins that are highly abundant without direct correlation to allergen exposure e.g. through plasma exudation. Moreover, the genomic and proteomic analysis could explain in more detail how the barrier of mucus and epithelium are affected by allergen exposure. The comparison to healthy controls and the longitudinal changes throughout the season further sheds light on how these individuals react upon allergen exposure and how this could lead to prevention of sensitization.

ELIGIBILITY:
Inclusion Criteria:

* pollen allergy verified by skin-prick test, blood tests for specific Immunoglobulin class E (RAST) and allergic rhinitis symptoms

Exclusion Criteria:

* chronic infectious diseases
* bad overall health condition
* malignant disease,
* pregnancy
* long-term intake of nasal and/or systemic steroids
* antihistamines or leukotrienes
* allergen immunotherapy
* acute and/or chronic rhinosinusitis
* parallel participation in other studies

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Allergic Rhinitis Patients and Healthy conrols
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Abundance Change of proteins | 1 year
  Abundance change of proteins will be measured semiquantitatively according to normalised mean areas under the curve of the respective experimental spectrum obtained from a distinct protein between the groups and seasons
Abundance Change of RNA/Genes | 1 year
  RNA Expression and gene expression will be measured by microarrays and fold changes will be obtained between the groups and seasons

CONTACTS AND LOCATIONS:
Locations (1):
- ENT University Hospital Graz, Graz, Styria, Austria